CLINICAL TRIAL: NCT01798459
Title: A Double Blind Randomized Crossover Study of the Effect of Methylphenidate Versus Placebo on State Anxiety in Children With Attention Deficit Hyperactivity Disorder.
Brief Title: The Effect of Methylphenidate Versus Placebo on State Anxiety in Children With Attention Deficit Hyperactivity Disorder.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Maya Kritchman Lupo, Resident, Shalvata Mental Health Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 0009-12-SHA
Record Dates: First submitted 2013-02-18; First posted 2013-02-25 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Methylphenidate; Placebo; State anxiety
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Anxiety Disorders | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Active Comparator): Methylphenidate 0.3 mg/kg per os is given before performing a continuous performance test.
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): Placebo is given before performing a continuous performance test.

INTERVENTIONS:
Drug: Methylphenidate
  Arms: Methylphenidate

SUMMARY:
The purpose of the study is to explore the effect of methylphenidate on state anxiety in children with attention deficit hyperactivity disorder.

Patient population: 30 children diagnosed with attention deficit hyperactivity disorder. The subjects will be of all racial, ethnical and gender categories, ranging from 8 to 18 years of age.

Structure: the study is a randomized double blind crossover study. The subjects will complete a continuous performance test, the cambridge neuropsychological test automated Battery, before and after given methylphenidate or placebo on the first day of the study. On the second day of the study, the subjects will receive either methylphenidate or placebo based on what was given on the first day of the study and they will complete the same task.

ELIGIBILITY:
Inclusion Criteria:

* Attention deficit and hyperactivity disorder
* Children aged 8-18 years

Exclusion Criteria:

* Pervasive developmental disorder
* Schizophrenia
* Bipolar disorder
* Current depressive episode
* Current Anxiety disorder
* Drug use during the past 6 months

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-10 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
State anxiety | 1 year
  State anxiety will be measured by the Spielberger's state anxiety inventory

SECONDARY OUTCOMES:
Cognitive function | 1 year
  Cognitive function will be measured by the cambridge neuropsychological test automated battery
Patient's perspective | 1 year
  Patient's perspective will be measured by questionnaires assessing treatment adherence issues and patient's view regarding the use of placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Kritchman Lupo, MD, Principal Investigator — Shalvata Mental Health Center
Locations (1):
- Shalvata, Hod HaSharon, Israel

REFERENCES:
- [Derived] Storebo OJ, Storm MRO, Pereira Ribeiro J, Skoog M, Groth C, Callesen HE, Schaug JP, Darling P, Huus CL, Zwi M, Kirubakaran R, Simonsen E, Gluud C. Methylphenidate for children and adolescents with attention deficit hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2025 Dec 4;12(12):CD009885. doi: 10.1002/14651858.CD009885.pub4. PMID 41342306
- [Derived] Storebo OJ, Storm MRO, Pereira Ribeiro J, Skoog M, Groth C, Callesen HE, Schaug JP, Darling Rasmussen P, Huus CL, Zwi M, Kirubakaran R, Simonsen E, Gluud C. Methylphenidate for children and adolescents with attention deficit hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD009885. doi: 10.1002/14651858.CD009885.pub3. PMID 36971690
- [Derived] Kritchman M, Koubi M, Mimouni Bloch A, Bloch Y. Effect of Methylphenidate on State Anxiety in Children With ADHD-A Single Dose, Placebo Controlled, Crossover Study. Front Behav Neurosci. 2019 May 15;13:106. doi: 10.3389/fnbeh.2019.00106. eCollection 2019. PMID 31156406